CLINICAL TRIAL: NCT07312357
Title: Electrostimulation Suit as a Therapeutic Tool in Post-COVID Syndrome: Effects on Physical and Functional Status. A Randomized Controlled Trial
Brief Title: Whole-Body Electrostimulation for Functional Recovery in Post-COVID Syndrome
Acronym: WB-EMS PostCOV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, María Del Pilar Rodríguez Pérez, Professor and Researcher, Department of Physiotherapy, Occupational Therapy, Rehabilitation and Physical Medicine, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A620-WBEMS-POSTCOVID; A620 (Other Grant/Funding Number: Universidad Rey Juan Carlos)
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Post COVID Syndrome Long Covid; Post COVID Syndrome; Long COVID Fatigue; Long Covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Whole-Body Electrostimulation (Experimental): Participants in this arm will receive active whole-body electromyostimulation using an electrostimulation suit during supervised functional activities. The intervention will consist of 12 weekly sessions with individualized and progressive stimulation parameters adjusted to achieve visible and tolerable muscle contractions.
  Interventions: Device: Whole-Body Electromyostimulation Suit
- Sham Whole-Body Electrostimulation (Placebo Comparator): Participants in this arm will use the same whole-body electrostimulation suit and perform the same supervised functional activities as the experimental group. The electrical stimulation will be set at minimal, non-therapeutic levels to act as a placebo condition, without expected physiological effects.
  Interventions: Device: Whole-Body Electromyostimulation Suit

INTERVENTIONS:
Device: Whole-Body Electromyostimulation Suit — The intervention consists of the use of a whole-body electromyostimulation (WB-EMS) suit with integrated surface electrodes designed to stimulate multiple large muscle groups simultaneously. Electrical stimulation is delivered at low-to-moderate frequencies and individualized intensities during supervised functional activities. Stimulation parameters are adjusted according to participant tolerance to achieve visible and tolerable muscle contractions. Sessions are conducted once per week for a total of 12 sessions, with progressive increases in session duration from 10 to 20 minutes. In the control condition, the same device is used with minimal, non-therapeutic electrical stimulation.

SUMMARY:
Post-COVID syndrome is a condition that affects some people after recovering from the acute phase of COVID-19. Common symptoms include persistent fatigue, reduced physical capacity, and difficulties performing everyday activities, which can significantly impact quality of life and independence. At present, there is limited scientific evidence on effective rehabilitation strategies for this population.

The purpose of this study is to evaluate whether the use of a whole-body electrostimulation suit can improve fatigue, physical performance, and functional independence in people with post-COVID syndrome. Whole-body electrostimulation is a non-pharmacological technique that uses low-frequency electrical impulses to activate multiple muscle groups simultaneously and has shown potential benefits in other clinical populations.

This is a randomized, double-blind, controlled pilot clinical trial. Participants will be randomly assigned to either an experimental group, which will receive active whole-body electrostimulation during functional activities, or a control group, which will follow the same sessions using the electrostimulation suit with minimal stimulation (placebo condition). Neither participants nor outcome assessors will know which group each participant belongs to.

The intervention will consist of 12 supervised sessions conducted once per week. Outcomes will be assessed before and after the intervention, with an additional follow-up assessment three months later. The main outcomes include fatigue levels, functional capacity, physical performance, and independence in activities of daily living. Safety and tolerance to the intervention will be monitored throughout the study.

The results of this study may help to determine the feasibility and potential effectiveness of whole-body electrostimulation as a rehabilitation tool for people with post-COVID syndrome and provide preliminary data for future larger-scale clinical trials.

DETAILED DESCRIPTION:
Post-COVID syndrome, also referred to as long COVID, is characterized by the persistence of physical, functional, and cognitive symptoms following acute SARS-CoV-2 infection. Fatigue, reduced exercise tolerance, and limitations in activities of daily living are among the most frequently reported and disabling symptoms. Despite the growing number of affected individuals, evidence-based rehabilitation strategies for this population remain limited.

Whole-body electromyostimulation (WB-EMS) is a non-pharmacological intervention that involves the simultaneous activation of large muscle groups through low-frequency electrical impulses delivered via surface electrodes integrated into a wearable suit. This technique allows muscle activation with low mechanical load and has shown potential benefits in improving physical performance and functional capacity in different clinical populations. However, its effectiveness in individuals with post-COVID syndrome has not yet been established.

This study is designed as a randomized, double-blind, controlled pilot clinical trial to evaluate the feasibility, safety, and preliminary effectiveness of a WB-EMS-based intervention in people with post-COVID syndrome. Participants will be randomly assigned to one of two groups: an experimental group receiving active WB-EMS during the performance of functional activities, and a control group undergoing the same intervention protocol with minimal electrical stimulation, intended to act as a placebo condition. Both participants and outcome assessors will be blinded to group allocation.

The intervention will consist of 12 supervised sessions, delivered once per week. Session duration will progressively increase from 10 to a maximum of 20 minutes, according to participant tolerance and protocol progression. Electrical stimulation parameters will be individualized and adjusted to achieve visible and tolerable muscle contractions in the experimental group, while remaining at non-therapeutic levels in the control group. Functional activities performed during the sessions will be selected and graded by qualified health professionals, with the aim of improving physical capacity, fatigue management, and independence in activities of daily living.

Outcome measures will be collected at baseline (pre-intervention), immediately after completion of the intervention (post-intervention), and at a three-month follow-up. Primary outcomes include fatigue and functional capacity. Secondary outcomes include physical performance, muscle strength, and independence in activities of daily living. Safety outcomes and adverse events will be monitored throughout the study.

As a pilot trial, this study aims to assess the feasibility and acceptability of the intervention, as well as to generate preliminary data on its potential therapeutic effects. The findings will inform the design of future larger-scale randomized controlled trials and contribute to the development of rehabilitation strategies for individuals with post-COVID syndrome.

ELIGIBILITY:
Inclusion Criteria:Adults aged 18 years or older.

Diagnosis of post-COVID syndrome (long COVID), with persistent symptoms following SARS-CoV-2 infection.

Presence of fatigue and/or functional limitations associated with post-COVID syndrome.

Ability to understand the study procedures and provide written informed consent.

Ability to participate in the intervention and assessments according to the study protocol.

-

Exclusion Criteria:

Participation in other structured physical exercise or rehabilitation programs during the study period.

Presence of severe cardiovascular disease or uncontrolled medical conditions that contraindicate physical activity or electrostimulation.

Neurological disorders or severe neuromuscular diseases.

Use of anabolic drugs or medications that may interfere with muscle function.

Pregnancy.

Epilepsy.

Active skin lesions or dermatological conditions in areas where electrodes are applied.

Recent oncological surgery.

Acute venous thrombosis.

Presence of cardiac pacemakers or implanted electronic or conductive medical devices.

Any clinical deterioration or condition that, in the opinion of the investigators, would make participation unsafe.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity | Baseline, immediately post-intervention (12 weeks), and 3-month follow-up
  Fatigue will be assessed using the Chalder Fatigue Scale (CFQ-11), a validated self-report questionnaire that evaluates physical and mental fatigue. Higher scores indicate greater fatigue severity.
Handgrip Muscle Strength | Baseline, immediately post-intervention (12 weeks), and 3-month follow-up
  Handgrip strength will be measured using a hand-held dynamometer as an objective indicator of overall muscle strength. Measurements will be performed following standardized procedures.

SECONDARY OUTCOMES:
Independence in Activities of Daily Living | Baseline, immediately post-intervention (12 weeks), and 3-month follow-up
  Independence in activities of daily living will be assessed using the Activities of Daily Living Questionnaire (ADLQ), a self-report instrument that evaluates functional independence across daily activities. Lower scores indicate greater functional independence.
Functional Capacity | Baseline, immediately post-intervention (12 weeks), and 3-month follow-up
  Functional capacity will be evaluated using the Six-Minute Walk Test (6MWT), which measures the maximum distance walked in six minutes as an indicator of aerobic capacity and functional exercise tolerance.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to data protection regulations and the sensitive nature of the health information collected.